CLINICAL TRIAL: NCT06724224
Title: Comparison of Levothyroxine Formulations in the Treatment of Congenital Hypothyroidism
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: TreatCHPed; 012/2024/Oss/AOUBo (Other: Comitato Etico Area Vasta Emilia Centro (CE-AVEC))
Record Dates: First submitted 2024-09-24; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-09

CONDITIONS: Congenital Hypothyroidism
MeSH Terms: conditions — Congenital Hypothyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Observational, retrospective, prospective, pharmacological, single-centre, non-profit study.

The aim is to evaluate, in newborns diagnosed with Congenital Hypothyroidism, the medium- and long-term efficacy and safety of the new formulation of levothyroxine in oral solution, compared to the liquid drop formulation and the tablet formulation.

The study will involve male and female patients referred to the Neonatal Screening Centre at the Centre for Endocrine-Metabolic Diseases of the Paediatrics Unit, IRCCS Azienda Ospedaliero-Universitaria di Bologna Policlinico di S. Orsola, Italy, who tested positive for Congenital Hypothyroidism.

DETAILED DESCRIPTION:
The prospective cohort consists of patients with Congenital Hypothyroidism identified through Neonatal Screening, who come for observation at the Centre for Endocrine-Metabolic Diseases of the Pediatrics Unit, IRCCS Azienda Ospedaliero-Universitaria di Bologna Policlinico di S. Orsola, Italy, from the approval of the study until the number of patients stipulated in the protocol is reached, which is expected to be achieved in about 4 years. The recruited patients will be assigned, based on the therapy taken in normal clinical practice, to a pharmacological group (group A: drops, group B: oral solution, group C: tablets), and their medical history, clinical and biochemical data will be collected at diagnosis.

The retrospective cohort includes children born from January 1, 2019 to the date of study approval, who came for observation at the Centre for Endocrine-Metabolic Diseases of the Pediatrics Unit, IRCCS Azienda Ospedaliero-Universitaria di Bologna Policlinico di S. Orsola, Italy, for Congenital Hypothyroidism identified by Neonatal Screening. These patients had levothyroxine therapy in one of the three formulations (solid, drops, oral solution) assigned according to normal clinical practice and will therefore be divided into 3 groups as for the prospective cohort. For these patients, retrospective collection and analysis of anamnestic, clinical, biochemical and radiological data and clinical, biochemical and neurocognitive follow-up is planned with the same timelines defined for the prospective cohort.

ELIGIBILITY:
Inclusion Criteria:

Newborn screening test positivity for Congenital Hypothyroidism; Subjects born in Emilia-Romagna region, Italy, and undergoing diagnostic confirmation and initiation of replacement therapy; Diagnosis-confirmed subjects who underwent L-T4 replacement therapy in the first month of life at Center for Endocrine-Metabolic Diseases, Pediatrics Units of the IRCCS Azienda Ospedaliero-Universitaria di Bologna Policlinico di S.Orsola, Italy; Age ≤11 years old; Obtaining informed consent from parents and/or legal guardians and assent from minors included in the study.

Exclusion Criteria:

Known chromosomal abnormalities or complex syndromes; Patients transferred to another center before completion of at least one year of follow-up from the start of therapy; Patients who started therapy at another center.

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients of both sex refer to the Neonatal Screening Center at the Center for Endocrine-Metabolic Diseases, Pediatrics Unit of the IRCCS Azienda Ospedaliero-Universitaria di Bologna Policlinico di S.Orsola, Italy, who test positive for Neonatal Screening for Congenital Hypothyroidism.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2031-04-08 (Estimated); Study Completion 2031-10-08 (Estimated)

PRIMARY OUTCOMES:
Mean and median values of TSH | at 7-15 days, at 1-3-6-12 months and thereafter annually until 3 years after the start of therapy
  microU/mL
Mean and median values of FT4 | at 7-15 days, at 1-3-6-12 months and thereafter annually until 3 years after the start of therapy
  pg/mL
Neuromotor-Neurocognitive development | at 1-3 years of age
  Griffiths Scale for patients aged 0-2 years; WPPSI-III Scale for patients aged 2.6-7.3 years
Proportion of patients with adverse effects | at 7-15 days, at 1-3-6-12 months and thereafter annually until 3 years after the start of therapy
  hypersensitivity reactions, tachycardia, irritability, headache, sweating, diarrhea, vomiting, heat intolerance

CONTACTS AND LOCATIONS:
Overall Officials: Rita Ortolano, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No